CLINICAL TRIAL: NCT01290289
Title: Analgesia in Labor, a Prospective Parallel Single Blind Study to Compare Regional Analgesia (Combined Spinal Epidural Analgesia (CSE), Epidural Analgesia (E)) and Intravenous (IV) Pethidine Analgesia
Brief Title: Analgesia in Labor, a Prospective Parallel Study to Compare Regional Analgesia and Intravenous (IV) Pethidine Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Nabila Sweed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6111972
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2009-07

CONDITIONS: Labor Active Dilated Cm
Keywords: Labor; Epidural; Combined spinal epidural; pethidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epidura, combined spinal epidura & IV (Active Comparator): Gp 1: received CSE analgesia, 25µg of fentanyl injected intrathecally & a bolus of 10 ml of 0.5% lidocaine injected epidurally.
  Gp 2: received CSE analgesia, 25µg of fentanyl injected intrathecally & a bolus of 10 ml of 0.0625% bupivacaine injected epidurally.
  Gp 3: received 50µg of E fentanyl analgesia, injected intrathecally & a bolus of 10 ml of 0.5% lidocaine, followed by lidocaine E top-ups.
  Gp 4: received 50µg of E fentanyl injected intrathecally and a bolus dose of 10 ml of 0.125% bupivacaine, followed by E bupivacaine top-ups.
  Gp 5: 50mg of IV pethidine was administered as a loading dose, followed by 0.5 mg/kg.
  Interventions: Other: Epidura, CSE & IV

INTERVENTIONS:
Other: Epidura, CSE & IV — Gp 1: received CSE analgesia: 25µg of fentanyl & a bolus dose of 10 ml of 0.5% lidocaine was injected epidurally. E top-ups of 5-10 ml of 0.5-0.8% lidocaine were then injected.
  Gp 2: received CSE analgesia: 25µg of fentanyl & a bolus dose of 10 ml of 0.0625% bupivacaine was injected epidurally. E top-ups of 5-10 ml of 0.0625-0.25% bupivacaine were then injected.
  Gp 3: received 50µg of E fentanyl analgesia & a bolus of 10 ml of 0.5% lidocaine was administered, followed by lidocaine E top-ups of 5-10 ml of 0.5-0.8%.
  Gp 4: received analgesia: 50µg of E fentanyl & a bolus dose of 10 ml of 0.125% bupivacaine was administered, followed by E bupivacaine top-ups of 5-10 ml of 0.125-0.25%.
  Gp 5: 50mg of IV pethidine was administered as loading dose, followed by 0.5 mg/kg.

SUMMARY:
To compare combined spinal epidural, epidural and IV pethidine analgesia and their effects on the mother, fetus, newborn and the course of labor.

DETAILED DESCRIPTION:
This is a prospective parallel single blind study, which was approved by the institutional review board of El-Galaa Teaching Hospital, and the research and ethics committee of Faculty of Pharmacy, Cairo University.

This hospital per si was selected for the study because it is large hospital that could provide the study with a diverse population. It has a population of various socio-economic statuses. This would provide the study with a sample of patients with a wide range of characteristics.

Sixty full-term, ASA physical status I or II nulliparous women in active labor with cervical dilatation of 5 cm and cephalic presenting fetus were randomly assigned to one of five groups after providing informed consent.

* Group 1: received CSE analgesia, where 25 µg of fentanyl was injected intrathecally and a bolus dose of 10 ml of 0.5% lidocaine was injected epidurally. E top-ups of 5-10 ml of 0.5-0.8% lidocaine were then injected upon request.
* Group 2: received CSE analgesia, where 25 µg of fentanyl was injected intrathecally and a bolus dose of 10 ml of 0.0625% bupivacaine was injected epidurally. E top-ups of 5-10 ml of 0.0625-0.25% bupivacaine were then injected upon request.
* Group 3: received 50µg of E fentanyl analgesia which was injected intrathecally and a bolus of 10 ml of 0.5% lidocaine was administered through the catheter, followed by lidocaine E top-ups of 5-10 ml of 0.5-0.8% upon request.
* Group 4: received analgesia, where 50 µg of E fentanyl were injected intrathecally and a bolus dose of 10 ml of 0.125% bupivacaine was administered through the catheter, followed by E bupivacaine top-ups of 5-10 ml of 0.125-0.25% upon request.
* Group 5: 50 mg of IV pethidine was administered as a loading dose, followed by 0.5 mg/kg, with a total maximum limit of 130 mg.

Study Subjects Excluding Criteria Patients who had diabetes mellitus, neurological disease, pre-eclampsia, or patients who had received parenteral analgesics or patients with contraindication to E or spinal analgesia, or patients with sensitivity to local anesthetics or opioids were excluded from the study.

Study Method All the recruited subjects were screened before the administration of any analgesia. Systolic and diastolic pressures, heart rate and peripheral oxygen saturation (SpO2) were monitored. Fetal heart rate (FHR) was monitored using an external cardiotocograph monitor (Partoconter NST Nihon Kohden).

For the E groups, the degree of motor block was assessed according to a modified Bromage scale (Grade I: free movement of legs and feet; Grade II: just able to flex knees with free movement of feet; Grade III: unable to flex knees, but with free movements of feet; Grade IV: unable to move legs or feet) before administration of E analgesia, 10 and 30 minutes after the first dose. The start of the analgesia was regarded as time 0. The duration of analgesia was taken as the time from the beginning of analgesic injection (time 0) to the time of request for additional analgesia.

The number of analgesic top-ups was recorded and the intervals between each top-up, in addition to the volume and concentration of the drug injected.

The Visual Analogue Pain Scale (VAS) (0 mm = no pain, 100 mm = worst pain imaginable) was measured before administration of analgesia, 10 and 30 minutes after administration of each analgesic dose until the delivery of the baby.

Maternal arterial pressures, heart rate, SpO2, and FHR were noted before the analgesia was given, and afterwards every 30 minutes until delivery.

Maternal temperature was recorded before starting the analgesic regimen and thereafter every hour till the end of labor. Fever was defined as temperature of ≥ 38˚C.

The duration of each stage of labor together with the mode of delivery were recorded.

The total volume of drug injected, total concentration of drug injected, 1-min and 5-min APGAR scores, weight of the neonate were recorded.

Any experienced drug related problem by any of the recruited subjects were recorded.

ELIGIBILITY:
Inclusion Criteria:

full-term, ASA physical status I or II nulliparous women in active labor with cervical dilatation of 5 cm and cephalic presenting fetus

Exclusion Criteria:

Patients who had diabetes mellitus, neurological disease, pre-eclampsia, or patients who had received parenteral analgesics or patients with contraindication to E or spinal analgesia, or patients with sensitivity to local anesthetics or opioids were excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale to assess pain control | 24 hours
  The Visual Analogue Pain Scale (VAS) (0 mm = no pain, 100 mm = worst pain imaginable) was measured before administration of analgesia, 10 and 30 minutes after administration of each analgesic dose until the delivery of the baby.

SECONDARY OUTCOMES:
The degree of motor block | 24 hours
  The degree of motor block was assessed according to a modified Bromage scale (Grade I: free movement of legs and feet; Grade II: just able to flex knees with free movement of feet; Grade III: unable to flex knees, but with free movements of feet; Grade IV: unable to move legs or feet) before administration of E analgesia, 10 and 30 minutes after the first dose. The start of the analgesia was regarded as time 0. The duration of analgesia was taken as the time from the beginning of analgesic injection (time 0) to the time of request for additional analgesia.
Number of top-ups | 24 hours
  The number of analgesic top-ups was recorded and the intervals between each top-up, in addition to the volume and concentration of the drug injected.
Adverse effects | 24 hours
  Any experienced drug related problem by any of the recruited subjects were recorded.
Labour Duration | 24 hours
  The duration of each stage of labor together with the mode of delivery were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nirmeen Sabry, Ph.D, Study Director — Cairo University
Locations (1):
- El-Galaa Hospital, Cairo, Egypt